CLINICAL TRIAL: NCT02471768
Title: The Association Between Central Aortic Blood Pressure Indices and Severity of Coronary Artery Disease
Acronym: CAPCAD
Status: Completed | Type: Observational
Sponsor: Government Medical College, Kozhikode (Other)
Responsible Party: Principal Investigator, SHREETAL RAJAN NAIR, Dr Shreetal Rajan Nair, Government Medical College, Kozhikode
Other Study IDs: Ref No IRC/2013/Protocol/162
Record Dates: First submitted 2015-06-08; First posted 2015-06-15 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease
Keywords: central pressure; Gensini score; pulsatility; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: CORONARY ANGIOGRAM AND CENTRAL AORTIC WAVEFORM ANALYSIS — coronary angiogram

SUMMARY:
Abstract

Objectives:

Primary: To study the association between central aortic blood pressure indices and coronary artery disease in patients undergoing elective angiography. Secondary: (a) To study whether any association exists between central aortic pressure indices and the incidence of major adverse cardiovascular events (MACE) in the same patients during a 6 month follow up period. (b) To study whether any association exists between the central aortic pressures and peripheral pressures.

Methods: The investigators conducted a prospective observational study in consecutive patients undergoing coronary angiography. Central and peripheral pressures were invasively recorded and coronary artery disease (CAD) classified into obstructive and non-obstructive group. CAD severity was graded using the Gensini score and subjects were divided into tertiles. Patients were followed up and the role of central aortic pressure indices in the prediction of cardiovascular events were analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective angiography for diagnosis of CAD.
* Age > 18 years

Exclusion Criteria:

* Patients with acute myocardial infarction, unstable angina or thromboembolism in the preceding 3 months.
* More than mild valvular heart disease.
* Renal impairment with serum creatinine > 1.5 mg%.
* Unable to obtain a full study of the coronary arteries.
* Peripheral vascular occlusive disease.
* Post coronary artery bypass grafting( CABG)
* Heart rate < 50/min and > 120/min and other arrhythmias.
* Contraindications for coronary angiography.
* Unable to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALL CONSECUTIVE SUBJECTS UNDERGOING CORONARY ANGIOGRAM FOR THE DIAGNOSIS OF CAD DURING A 6 MONTH PERIOD
Sampling Method: Probability Sample
Enrollment: 623 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
acute coronary syndrome(ACS) | 6 MONTHS
stroke | 6 months
revascularisation | 6 months
death | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: SHREETAL R NAIR, Principal Investigator — Government Medical College, Kozhikode